CLINICAL TRIAL: NCT04935775
Title: The Effect of Touch on Pain and Anxiety During the Bone Marrow Biopsy Procedure
Acronym: Dixon Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Anna D. Schaal, Hematology Nurse Practitioner, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: D21039
Record Dates: First submitted 2021-06-02; First posted 2021-06-23 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Pain, Acute; Anxiety
MeSH Terms: conditions — Acute Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Untrained Touch Provided (Experimental)
  Interventions: Other: Untrained Touch
- Standard of Care (No Intervention)

INTERVENTIONS:
Other: Untrained Touch — Subject's feet, ankles, and lower legs are touched and rubbed during a bone marrow biopsy procedure.
  Arms: Untrained Touch Provided

SUMMARY:
This study is analyzing the benefit of untrained touch provided during a bone marrow biopsy procedure as compared to performing the procedure without providing it.

DETAILED DESCRIPTION:
Two protocol-identified licensed nursing aides (LNA) will provide an unstructured simple touch intervention that requires no special training other than being oriented to "rub patient's feet" during the procedure. Data will be collected through patient-reported outcomes to determine if "untrained" touch has therapeutic results in managing a patient's pain and anxiety during a bone marrow biopsy procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients from Norris Cotton Cancer Center who have been scheduled for a bone marrow biopsy at the Outpatient Surgical Center at Dartmouth-Hitchcock Medical Center.
2. Subjects must be able to read and write in English to provide informed consent and fill out the questionnaires.

Exclusion Criteria:

1. Patients who do not wish to have their feet and lower legs touched during the procedure
2. Open sores on their feet or lower legs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Evaluate patient-reported pain levels | During the study procedure
  Patients be asked to describe what their pain level was before, at its worst point during the procedure and after the bone marrow biopsy. The Visual Analog Scale (VAS) will be used on a 0 to 10 scale, 0 being no pain at all and 10 being the worst pain imaginable.
Evaluate patient-reported anxiety levels | During the study procedure
  The six -item short form Spiellberger State-Trait Anxiety Inventory (STAI), a self-reported questionnaire, will be administered on pencil and paper. Possible ranges of scores on the 6-item questionnaires vary from 6 to 24, with separate scores for both the state and trait anxiety sections. Answers to each question range from 1 to 4, 1 being no anxiety at all to 4 being very high anxiety (Julian, 2014). Patients will complete the short-form STAI before and after the procedure.
Identify correlation between demographics and interventional response | During the study procedure
  Secondary endpoints will include identifying any correlation between demographic data collected and response to the intervention. The patient experience will be evaluated by using a visual analog scale at the completion of the procedure via paper and pencil that the subjects will complete independently. These open ended questions will be used to inform larger study questions in the future. Abstracted and deidentified summaries of responses will be prepared by the study PI.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Schaal, MSN, APRN, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Dartmouth Cancer Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baldwin AL, Vitale A, Brownell E, Kryak E, Rand W. Effects of Reiki on Pain, Anxiety, and Blood Pressure in Patients Undergoing Knee Replacement: A Pilot Study. Holist Nurs Pract. 2017 Mar/Apr;31(2):80-89. doi: 10.1097/HNP.0000000000000195. PMID 28181973
- [Background] Abdelaziz, S. H., & Mohammed, H. E. (2014). Effect of foot massage on postoperative pain and vital signs in breast cancer patient. Journal of Nursing Education and Practice, 4(8). doi:10.5430/jnep.v4n8p115
- [Background] Bao T, Ye X, Skinner J, Cao B, Fisher J, Nesbit S, Grossman SA. The analgesic effect of magnetic acupressure in cancer patients undergoing bone marrow aspiration and biopsy: a randomized, blinded, controlled trial. J Pain Symptom Manage. 2011 Jun;41(6):995-1002. doi: 10.1016/j.jpainsymman.2010.08.012. Epub 2011 Feb 9. PMID 21306863
- [Background] Birocco N, Guillame C, Storto S, Ritorto G, Catino C, Gir N, Balestra L, Tealdi G, Orecchia C, Vito GD, Giaretto L, Donadio M, Bertetto O, Schena M, Ciuffreda L. The effects of Reiki therapy on pain and anxiety in patients attending a day oncology and infusion services unit. Am J Hosp Palliat Care. 2012 Jun;29(4):290-4. doi: 10.1177/1049909111420859. Epub 2011 Oct 13. PMID 21998438
- [Background] Bourque AL, Sullivan ME, Winter MR. Reiki as a pain management adjunct in screening colonoscopy. Gastroenterol Nurs. 2012 Sep;35(5):308-12. doi: 10.1097/SGA.0b013e3182603436. PMID 23018166
- [Background] Brunetti GA, Tendas A, Meloni E, Mancini D, Maggiore P, Scaramucci L, Giovannini M, Niscola P, Cartoni C, Alimena G. Pain and anxiety associated with bone marrow aspiration and biopsy: a prospective study on 152 Italian patients with hematological malignancies. Ann Hematol. 2011 Oct;90(10):1233-5. doi: 10.1007/s00277-011-1166-7. Epub 2011 Feb 2. No abstract available. PMID 21287348
- [Background] Ferrell-Torry AT, Glick OJ. The use of therapeutic massage as a nursing intervention to modify anxiety and the perception of cancer pain. Cancer Nurs. 1993 Apr;16(2):93-101. PMID 8477405
- [Background] Gay CW, Robinson ME, George SZ, Perlstein WM, Bishop MD. Immediate changes after manual therapy in resting-state functional connectivity as measured by functional magnetic resonance imaging in participants with induced low back pain. J Manipulative Physiol Ther. 2014 Nov-Dec;37(9):614-27. doi: 10.1016/j.jmpt.2014.09.001. Epub 2014 Oct 3. PMID 25284739
- [Background] Gonella S, Garrino L, Dimonte V. Biofield therapies and cancer-related symptoms: a review. Clin J Oncol Nurs. 2014 Oct;18(5):568-76. doi: 10.1188/14.CJON.568-576. PMID 25253110
- [Background] Gorji, A., Taebei, M., Ranjbar, M., & Hatkehlouei, M. (2016). Effect of Distraction Technique and Hypnosis in Pain of Bone Marrow Aspiration in Children: A Systematic Review Study. International Journal of Pediatrics, 5(3). doi:10.22038/ijp.2016.20976.1754
- [Background] Grealish L, Lomasney A, Whiteman B. Foot massage. A nursing intervention to modify the distressing symptoms of pain and nausea in patients hospitalized with cancer. Cancer Nurs. 2000 Jun;23(3):237-43. doi: 10.1097/00002820-200006000-00012. PMID 10851775
- [Background] Hart LK, Freel MI, Haylock PJ, Lutgendorf SK. The use of healing touch in integrative oncology. Clin J Oncol Nurs. 2011 Oct;15(5):519-25. doi: 10.1188/11.CJON.519-525. PMID 21951738
- [Background] Hjortholm N, Jaddini E, Halaburda K, Snarski E. Strategies of pain reduction during the bone marrow biopsy. Ann Hematol. 2013 Jan;92(2):145-9. doi: 10.1007/s00277-012-1641-9. Epub 2012 Dec 6. PMID 23224244
- [Background] Johnson H, Burke D, Plews C, Newell R, Parapia L. Improving the patient's experience of a bone marrow biopsy - an RCT. J Clin Nurs. 2008 Mar;17(6):717-25. doi: 10.1111/j.1365-2702.2007.01991.x. Epub 2007 Nov 30. PMID 18047576
- [Background] Kuball, J., Shuz, J., Gamm, H., & Weber, M. (n.d.). Bone marrow punctures and pain. Acute Pain, 6(1), 9-14. doi:10.1016/j.acpain.2004.02.003
- [Background] Kutner JS, Smith MC, Corbin L, Hemphill L, Benton K, Mellis BK, Beaty B, Felton S, Yamashita TE, Bryant LL, Fairclough DL. Massage therapy versus simple touch to improve pain and mood in patients with advanced cancer: a randomized trial. Ann Intern Med. 2008 Sep 16;149(6):369-79. doi: 10.7326/0003-4819-149-6-200809160-00003. PMID 18794556
- [Background] Lutgendorf SK, Mullen-Houser E, Russell D, Degeest K, Jacobson G, Hart L, Bender D, Anderson B, Buekers TE, Goodheart MJ, Antoni MH, Sood AK, Lubaroff DM. Preservation of immune function in cervical cancer patients during chemoradiation using a novel integrative approach. Brain Behav Immun. 2010 Nov;24(8):1231-40. doi: 10.1016/j.bbi.2010.06.014. Epub 2010 Jun 30. PMID 20600809
- [Background] Robison JG, Smith CL. Therapeutic Massage During Chemotherapy and/or Biotherapy Infusions: Patient Perceptions of Pain, Fatigue, Nausea, Anxiety, and Satisfaction. Clin J Oncol Nurs. 2016 Apr;20(2):E34-40. doi: 10.1188/16.CJON.E34-E40. PMID 26991721
- [Background] Rosenbaum MS, Velde J. The Effects of Yoga, Massage, and Reiki on Patient Well-Being at a Cancer Resource Center. Clin J Oncol Nurs. 2016 Jun 1;20(3):E77-81. doi: 10.1188/16.CJON.E77-E81. PMID 27206308
- [Background] Snow A, Dorfman D, Warbet R, Cammarata M, Eisenman S, Zilberfein F, Isola L, Navada S. A randomized trial of hypnosis for relief of pain and anxiety in adult cancer patients undergoing bone marrow procedures. J Psychosoc Oncol. 2012;30(3):281-93. doi: 10.1080/07347332.2012.664261. PMID 22571244
- [Background] Jane SW, Wilkie DJ, Gallucci BB, Beaton RD. Systematic review of massage intervention for adult patients with cancer: a methodological perspective. Cancer Nurs. 2008 Nov-Dec;31(6):E24-35. doi: 10.1097/01.NCC.0000339242.51291.85. PMID 18987505
- [Background] Tabatabaee A, Tafreshi MZ, Rassouli M, Aledavood SA, AlaviMajd H, Farahmand SK. EFFECT OF THERAPEUTIC TOUCH ON PAIN RELATED PARAMETERS IN PATIENTS WITH CANCER: A RANDOMIZED CLINICAL TRIAL. Mater Sociomed. 2016 Jun;28(3):220-3. doi: 10.5455/msm.2016.28.220-223. Epub 2016 Jun 1. PMID 27482166
- [Background] Thrane S, Cohen SM. Effect of Reiki therapy on pain and anxiety in adults: an in-depth literature review of randomized trials with effect size calculations. Pain Manag Nurs. 2014 Dec;15(4):897-908. doi: 10.1016/j.pmn.2013.07.008. Epub 2014 Feb 28. PMID 24582620
- [Background] Tucker DL, Rockett M, Hasan M, Poplar S, Rule SA. Does transcutaneous electrical nerve stimulation (TENS) alleviate the pain experienced during bone marrow sampling in addition to standard techniques? A randomised, double-blinded, controlled trial. J Clin Pathol. 2015 Jun;68(6):479-83. doi: 10.1136/jclinpath-2015-202908. Epub 2015 Mar 10. PMID 25759407
- [Background] Ucuzal M, Kanan N. Foot massage: effectiveness on postoperative pain in breast surgery patients. Pain Manag Nurs. 2014 Jun;15(2):458-65. doi: 10.1016/j.pmn.2012.03.001. Epub 2012 Jun 20. PMID 24882025
- [Background] Watmough S, Flynn M. A review of pain management interventions in bone marrow biopsy. J Clin Nurs. 2011 Mar;20(5-6):615-23. doi: 10.1111/j.1365-2702.2010.03485.x. PMID 21320190
- [Background] Weze C, Leathard HL, Grange J, Tiplady P, Stevens G. Evaluation of healing by gentle touch in 35 clients with cancer. Eur J Oncol Nurs. 2004 Mar;8(1):40-9. doi: 10.1016/j.ejon.2003.10.004. PMID 15003743